CLINICAL TRIAL: NCT01708811
Title: Will Reduction in Plasma Sodium Reduce Myometrium Contractility in Humans? An Invitro Study of Pregnant Myometrium at Term.
Brief Title: Hyponatremia and Myometrium Contractility. An Invitro Study
Status: Terminated | Type: Observational
Why Stopped: Few biopsies showed the expected pattern We suspect erroeneous method.
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Moen, research fellow, Karolinska Institutet
Other Study IDs: LOF-KS1
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Hyponatremia
Keywords: Contractility; human; myometrium; hyponatraemia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biopsies of pregant myometrium
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyponatremia during labour has been associated with prolonged labour, and increased incidence of instrumental delivery and emergency caesarean section. Sodium influx in myometral cells are involved in contractility,and and influence of hyponatraemia on contractility can be suspected.

DETAILED DESCRIPTION:
Biopsies will be obtained from pregnant women undergoing planned caesarean section at term. The biopsies will divided into 3 strips that will be stored overnight in chilled NaCl 0.9%. The following morning each strip will be mounted isometrically with one end fixed to a holder and the other end to a force transducer. One strip will be maintained in a solution containing 140mmol/L Na,acting as control, whereas the other two strips will be placed in fluids with diminishing Na concentration, from 140 mmol/L, to 130 mmol/L and 120 mmol/L. Contractility will be measured with force transducers and a polygraph

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at term

Exclusion Criteria:

* Preeclampsia

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy women with singleton pregancies requiring delivery planned caesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Contractility | 24 hours
  Contractility will be measured, and data analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Gunvor Ekman-Ordeberg, PhD, Principal Investigator — Department of Women and Child´s Healt, karolinska University Hospital, Solna, Stockholm, Sweden
Locations (1):
- Department of Women and Child´s Health, Karolinska University Hospital, Solna, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Moen V, Brudin L, Rundgren M, Irestedt L. Hyponatremia complicating labour--rare or unrecognised? A prospective observational study. BJOG. 2009 Mar;116(4):552-61. doi: 10.1111/j.1471-0528.2008.02063.x. Epub 2009 Jan 27. PMID 19175600
- [Background] Kamizaki J, Shimizu K, Nakajyo S, Urakawa N. A comparative study on the contraction induced by high K+/Na+ deficient solution in rat uterus or urinary bladder. Jpn J Pharmacol. 1988 Jun;47(2):179-88. doi: 10.1254/jjp.47.179. PMID 3199594
- [Background] Sperelakis N, Inoue Y, Ohya Y. Fast Na+ channels and slow Ca2+ current in smooth muscle from pregnant rat uterus. Mol Cell Biochem. 1992 Sep 8;114(1-2):79-89. PMID 1281264
- [Background] Cheek TG, Samuels P, Miller F, Tobin M, Gutsche BB. Normal saline i.v. fluid load decreases uterine activity in active labour. Br J Anaesth. 1996 Nov;77(5):632-5. doi: 10.1093/bja/77.5.632. PMID 8957980
- [Background] Garite TJ, Weeks J, Peters-Phair K, Pattillo C, Brewster WR. A randomized controlled trial of the effect of increased intravenous hydration on the course of labor in nulliparous women. Am J Obstet Gynecol. 2000 Dec;183(6):1544-8. doi: 10.1067/mob.2000.107884. PMID 11120525